CLINICAL TRIAL: NCT01687491
Title: Comparison of Anti-Xa Activity in the Treatment With Enoxaparin in ACS Admitted to the Emergency. Randomized Clinical Trial ENOXA ® Versus LOVENOX ®
Brief Title: Comparison of Anti-Xa Activity of ENOXA ® Versus LOVENOX ® in Acute Coronary Syndrome
Acronym: AXA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Collaborators: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AXA_2012
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2012-09

CONDITIONS: Acute Coronary Syndrome; Factor X
Keywords: Enoxaparin; Acute Coronary Syndrome; Factor X
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enoxa (Active Comparator): ENOXA® Anti-Xa/kg 100 IU by subcutaneous injection every 12 hours
  Interventions: Drug: ENOXA®
- Lovenox (Active Comparator): LOVENOX® Anti-Xa/kg 100 IU by subcutaneous injection every 12 hours
  Interventions: Drug: LOVENOX®

INTERVENTIONS:
Drug: ENOXA® — enoxaparine 100 UI/Kg subcutaneous injection
  Arms: Enoxa
Drug: LOVENOX® — enoxaparine 100 UI/Kg subcutaneous injection
  Arms: Lovenox

SUMMARY:
This study is a clinical trial monocentric, open, randomized ENOXA ® versus LOVENOX ®, conducted on two parallel groups of patients admitted in emergency for acute coronary syndrome.

DETAILED DESCRIPTION:
The patients included in this study with an acute coronary Syndrome be admitted to the emergency room and receive treatment with enoxaparin. Low molecular weight heparin (LMWH) treatment in this indication is usually spread over a week. The experience of the study intends to focus only on the first injection administered in selected patients.

Two assays are carried out, including an assessment of the anti-Xa activity initially before injection of enoxaparin, and 4 hours after administration of the first syringe.

Clinical monitoring is intrahospital from the date of hospitalization of patients included until emergency exit (transfer to another service, or return home)

Tolerance assessment (clinical and biological) is performed during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 20 years
* acute coronary syndrome
* Admission to the emergency department

Exclusion Criteria:

* Patient participating in another study
* Pregnant or lactating or of childbearing potential not using medically accepted method of contraception
* Taking an anticoagulant in the last three months
* Patient with known haemostatic disorder
* Contraindication absolute and / or relative to the use of enoxaparin
* Nobody wishing to participate in this study or not having the ability to understand its objectives

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
anti-Xa activity | 4 hours
  assay of anti-Xa activity 4 hours after the first injection énoxparine

SECONDARY OUTCOMES:
adverse events | participants will be followed for the duration of hospital stay, an expected average of 7 days
  Tolerance is assessed by the occurrence of adverse events and / or serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, PHD, Study Chair — Fattouma Bourguiba Hospital, Monastir; Mohsen Hassine, Principal Investigator — Fattouma Bourguiba, Monastir
Locations (1):
- Departement of Emergency, Monastir, Monastir Governorate, Tunisia

REFERENCES:
- [Background] Boubaker H MD, Grissa MH MD, Sassi M MD, Chakroun T MD, Beltaief K MD, et al. (2015) Generic and Branded Enoxaparin Bioequivalence: A Clinical and Experimental Study. J Bioequiv Availab 7: 225-228. doi:10.4172/jbb.1000244
- See also: abstract link posted on the journal's website — http://www.omicsonline.org/bioequivalence-bioavailability-abstract.php?abstract_id=56339
- See also: PDF full text of article published on Journal of Bioequivalence & Bioavailability (open access) — http://www.omicsonline.org/open-access/generic-and-branded-enoxaparin-bioequivalence-a-clinical-andexperimental-study-jbb-1000244.pdf